CLINICAL TRIAL: NCT05875714
Title: Apremilast for the Treatment of Refractory Erythema Multiforme
Brief Title: Apremilast for Erythema Multiforme
Acronym: AEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Micheletti (Other)
Responsible Party: Sponsor-Investigator, Robert Micheletti, Associate Professor of Dermatology and Medicine, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 842831
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Erythema Multiforme
MeSH Terms: conditions — Erythema Multiforme | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Apremilast — Apremilast (Otezla), oral medication Day 1: 10 mg in the morning. Day 2: 10 mg in the morning and 10 mg in the evening. Day 3: 10 mg in the morning and 20 mg in the evening. Day 4: 20 mg in the morning and 20 mg in the evening. Day 5: 20 mg in the morning and 30 mg in the evening Day 6: 30 mg twice daily Maintenance dosing: 30 mg twice daily
  Other Names: Otezla

SUMMARY:
This study is recruiting patients with chronic, treatment resistant erythema multiforme (EM), which is a disease that can affect the skin and mucous membranes (mucocutaneous). EM often impacts quality of life with pain, anorexia, hospitalization, and related long-term issues. While there are medications used to treat EM, no single therapeutic agent has been consistently effective for long-term management of disease. Apremilast (trade name: Otezla) is approved to treat Bechet's Disease, a different but similar mucocutaneous disease. In this study, eligible patients will receive apremilast for 6 months of treatment so we can evaluate if there is a difference in pain and the number of EM flares compared to prior to treatment with apremilast.

ELIGIBILITY:
Inclusion Criteria

Subjects must satisfy the following criteria to be enrolled in the study:

1. Presence of oral, genital, or cutaneous erythema multiforme (EM) diagnosed or confirmed by a dermatologist based on clinical and/or histopathologic data.
2. EM must be recurrent, defined as having =>2 flares in the six months prior to enrollment (or =>4 flares in the year prior to enrollment).
3. EM must be refractory to standard therapy defined as 3-month treatment course with valacyclovir and/or a systemic immunomodulatory therapy such as colchicine, dapsone, azathioprine, mycophenolate mofetil, or methotrexate.
4. Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, and clinical laboratories. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
5. Willing and able to provide personally signed and dated informed consent form.
6. Stated willingness and ability to comply with all study procedures including adhering to oral apremilast regimen and availability for the duration of the study.
7. Adults aged 18-89 years old.
8. People of childbearing potential (PCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, PCBP who engage in activity by which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: External or internal condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

NOTE: This criterion is satisfied as "not applicable" (N/A) for those who practice abstinence as part of their usual and customary way of life, so long as this is maintained throughout study period plus 28 days post-treatment; are postmenopausal; or are of male sex/assigned male at birth (AMAB).

Exclusion Criteria

The presence of any of the following will exclude a subject from enrollment:

1. Other than disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinological, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
2. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if they were to participate in the study.
3. Prior history of unmanaged depressive symptoms, suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
4. A score of 4 or higher on Patient Health Questionnaire at screening.
5. Pregnant or breast feeding.
6. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
7. Malignancy or history of malignancy, except for:

   1. treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
   2. treated [ie, cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
8. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
9. Prior treatment with apremilast.
10. Patient unable to comply with study or conform to treatment diary or regular follow up visits.
11. Patients with ocular EM.
12. Concomitant use of immunosuppressive medications for treatment of other diseases.
13. Patients with contraindications to Apremilast according to package insert.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
EM flares on medication | 24 weeks
  Change in frequency and duration of EM flares at 24-week evaluation.

SECONDARY OUTCOMES:
Pain on medication | 24 weeks
  Change in pain severity (on 0 to 10 scale) of EM flares at 24-week evaluation
Flares off medication | 36 weeks
  Change in frequency and duration of flares at 36-week follow-up.
Pain off medication | 36 weeks
  Change in pain severity (on 0-10 visual analogue scale) of EM flares at 36-week follow-up.
Prednisone | 36 weeks
  Use of prednisone as rescue therapy to treat flares.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Micheletti, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center For Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No